CLINICAL TRIAL: NCT02954718
Title: Effects of Video-Based Task Oriented Activity Training on Activity Performance and Participation in Patients With Juvenile Idiopathic Arthritis
Brief Title: Video-Based Task Oriented Activity Training in Patients With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Saime Nilay Arman, Principal investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41260
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2015-02

CONDITIONS: Video-based Task Oriented Activity Training
Keywords: activity performance; juvenile idiopathic arthritis; virtual reality
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): patient-centered task oriented activity training in real life
  Interventions: Other: activity training
- 2 (Experimental): patient-centered video-based task oriented activity training
  Interventions: Other: activity training

INTERVENTIONS:
Other: activity training
  Other Names: exercise training

SUMMARY:
Juvenile idiopathic arthritis (JIA) is most common chronic rheumatic disease in childhood. The upper extremity involvement in JIA causes muscle imbalance, joint destruction, pain, stiffness and limitations on daily living activities (DLA) in varying degrees. However, the information about prevalence of symptoms, disorders, DLA limitations, participation restriction and options of treatments for upper extremity involvement in JIA are limited. It has been reported that improvements of upper extremity functions were achieved by video-based games (VBG) in various disease groups. However, in the literature, no study has been found about effectiveness of WBG in children with arthritis. The aim of the study was to investigate effects of task-oriented activity training (TOAT) with VBG versus activity training in real life on activity performance and participation in children with arthritis. Participants with upper limb involvement in JIA were randomly assigned to the activity training in real life group (group I) and TOAT with VBG in real life group (group II). The actual materials and rehabilitation kits will be used for activity training in group 1, the DLA that expected to gain independence will be trained with VBG in group 2. Upper extremity muscle strength and grip, range of motion, upper limb functions, activity, participation and quality of life will be evaluated. The hypothesis of this study is that TOAT with VBG improves the activity performance and physical functions and increases the participation, via being stimulative and interactive in order to provide feedback and to increase interest and motivation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as JIA according to ILAR classification
* Aged between 6-18
* At least one affected joint in upper extremity (shoulder, elbow, wrist, and hand joints)
* Adequate cognitive function in the compliance of exercise program

Exclusion Criteria:

• Surgery or arthroscopic operation in the last year

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Childhood Health Assessment Questionaire (CHAQ) | 8 weeks
Canadian Occupational Performance Measure (COPM) | 8 weeks

SECONDARY OUTCOMES:
Duruoz Hand Index | 8 weeks
Jebsen-Taylor Hand Function Test (JTHFT) | 8 weeks

REFERENCES:
- [Derived] Arman N, Tarakci E, Tarakci D, Kasapcopur O. Effects of Video Games-Based Task-Oriented Activity Training (Xbox 360 Kinect) on Activity Performance and Participation in Patients With Juvenile Idiopathic Arthritis: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2019 Mar;98(3):174-181. doi: 10.1097/PHM.0000000000001001. PMID 30020092